CLINICAL TRIAL: NCT00445510
Title: A Double Blind, Placebo Controlled, Repeat Dose Study to Determine the Effect of GSK256066 87.5 Mcg to Protect Against AMP Challenge in the Lung in Mild Steroid-naive Asthmatics.
Brief Title: This Study Will Examine the Effects of GSK256066 to Protect Mild Steroid-naive Asthmatics Against an Antigen Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IPA106620
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Asthma
Keywords: GSK256066,; allergen,; challenge,; repeat dose,; AMP,; mild asthmatics
MeSH Terms: conditions — Asthma | interventions — 6-((3-((dimethylamino)carbonyl)phenyl)sulfonyl)-8-methyl-4-((3-methyloxyphenyl)amino)-3-quinolinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK256066

SUMMARY:
This will be a single centre, randomised, double-blind, placebo-controlled, 2-period crossover study to investigate the effect of treatment with repeat inhaled doses of GSK256066 on bronchial hyper-reactivity to adenosine monophosphate.

ELIGIBILITY:
Inclusion: (All must Apply)

* Males and females aged 18 to 55 years inclusive.
* Documented history of bronchial asthma, first diagnosed at least 6 months prior to the screening visit and currently being treated only with intermittent short-acting beta -agonist therapy by inhalation.
* Pre-bronchodilator FEV1 >75% of predicted at screening.
* Documented sensitivity to AMP with a provocative concentration of AMP resulting in a 20% fall in FEV1 (PC20 AMP) of <80 mg/ml at the screening visit.
* Demonstrate stable bronchoconstriction in response to inhaled AMP at the run-in visit. 'Stable bronchoconstriction' is a term to define a population of asthmatics who have a repeatable and reproducible response to a challenge agent that induces bronchoconstriction. The run-in PC20 needs to be within 1.25DD of the screening PC20.
* Non-smoking status as verified by urinary cotinine levels below 300 ng/mL cotinine at the screening visit. This can include ex-smokers who have given up smoking for >6 months and have less than a 5 pack-year smoking history.
* Able and willing to give written informed consent to take part in the study.
* Available to complete all study measurements.

Exclusion:

* Pregnant or nursing females.
* Past or present disease, which as judged by the investigator, may affect the outcome of this study.
* Subject has known history of hypertension or is hypertensive at screening.
* Respiratory tract infection and/or exacerbation of asthma within 4 weeks prior to the first dose of study medication.
* History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnoea, respiratory arrest and/or hypoxic seizures.
* Unable to abstain from prescription medication, other than short acting inhaled beta-agonists and paracetamol for the treatment of minor ailments eg headache from 48h before the first dose until the follow-up visit.
* The subject has participated in a clinical trial during the previous 3 months.
* History of blood donation (450 mL) within 2 months of starting the clinical study.
* The subject regularly drinks more than 28 units of alcohol in a week if male, or 21 units per week if female.
* The subject has tested positive for hepatitis C antibody or hepatitis B surface antigen or HIV antibodies.
* The subject has positive drugs of abuse test.
* Subjects weighing less than 50kg are to be excluded from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24
Dates: Start 2006-06

PRIMARY OUTCOMES:
AMP PC20: GSK256066 7 days of 87.5mcg vs placebo 2hrs post-dose on Day 7.

SECONDARY OUTCOMES:
AMP PC20: GSK256066 7 days of 87.5mcg vs placebo 24hrs post-dose on Day 7. Exhaled Nitric Oxide: GSK256066 7 days of 87.5mcg vs placebo at Day 1; 1hr and 2hr, Day 7; 1hr, 2hr and 24hr.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wellington, New Zealand